CLINICAL TRIAL: NCT01727011
Title: A Phase I-II Trial Evaluating the Toxicity of Early Breast Partial Irradiation in Patients Aged at Least of 70 Years With Breast Cancer at Low Risk of Local Recurrence
Brief Title: Single Fraction Elderly Breast Irradiation (SiFEBI)
Acronym: SIFEBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/09 - SIFEBI; 2012-A00745-38 (Registry Identifier: 2012-A00745-38)
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Single fraction; Elderly; Breast Irradiation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IPAS (Experimental): Once the patient recorded in the trial, and after completion of a post-implant dosimetry scanner to analyze the dose distribution within the target volume and organs at risk, the patient is treated by irradiation and partial accelerated breast brachytherapy using high dose rate, delivering a total dose of 16 Gy in one fraction
  Interventions: Radiation: IPAS

INTERVENTIONS:
Radiation: IPAS
  Other Names: irradiation and partial accelerated breast brachytherapy

SUMMARY:
Irradiation and Accelerated Partial Breast (IPAS) to this day remains a therapeutic concept whose validity is being assessed on its non-inferiority in terms of local control compared to whole breast irradiation. At least eight phase III trials attempting to answer this question and thus provide a sufficient level of evidence to make this concept a new standard of care for sub-groups of patients well defined (1).

However, without waiting for the final results of these randomized trials (which will not be fully valid with a drop of at least ten years), the American societies (ASTRO) and European (ESTRO) radiotherapy have all two proposed classification (very similar) into 3 groups according to the risk to the patient in terms of local recurrence after IPAS. And are defined by the ESTRO:

* The low-risk group ("suitable" for ASTRO)
* The intermediate-risk group ("cautionary" in ASTRO)
* The high-risk group ("not suitable" for ASTRO) (2.3). Therefore, it is possible to propose to a patient a randomized clinical tria IPAS, to subject it belongs to the group "low risk." The results of phase II trials as a long-term analysis of the matched team of William Beaumont Hospital (4) and the phase III trial using intra-operative radiation photons in low energy X whose results were recently published (5) confirm the value of this new therapeutic concept for post-operative breast cancer at low risk of local recurrence.

In France, the therapists were quickly directed to a sub-population for which the IPAS could represent a real improvement in the therapeutic management in significantly reducing the number of irradiation sessions of thirty in 6 weeks 5 days at 10 in a single view (6). Several French phase II trials were started specifically targeting the female population aged using a balloon catheter (MammoSite ®) (7) or by intra-operative radiation électronthérapie (8). The results of the test using the GERICO-03 brachytherapy with high dose rate (promoter: FNCLCC, National Federation of Anti Cancer Centres , recently merged into Group Health Cooperation entitled UNICANCER) are currently submitted to Journal Green Radiotherapy (Radiotherapy and Oncology from 09/11/11) (9).

On a technical level, two main approaches are used (10):

* Irradiation intraoperative electron or low-energy photons,
* Radiation after surgery The advantage of intraoperative irradiation is the optimal reduction of total processing time radio-surgery because the patient is irradiated during the lumpectomy. However, 15-20% of these patients receive partial breast irradiation, as histo-prognostic criteria provided in the histologically final report, confirm the non-adapted indication of IPAS (5).

In contrast, the post-operative IPAS can treat only patients meeting all criteria for IPAS but treatment-related travel are about 5 treatments for bi-fractionated (2 sessions per days separated by at least 6 hours).

DETAILED DESCRIPTION:
Single dose intraoperative issued by electrontherapy or low energy photons (50 Kv) is 21 Gy (5.11). However, these doses reported in the irradiated volume are not equivalent. Indeed, with electrontherapy, it is a complete volume of mammary parenchyma that is irradiated, whereas with low energy photon therapy (X 50 KV) is a "shell" of 5 mm thick which is treated knowing that to 10 mm from the surface of the sphere of treatment, the gland received only 50% of the dose initially prescribed. On interstitial brachytherapy with high dose rate, it has a dose escalation due to intrinsic volumes located within the irradiated area that will receive a higher dose than prescribed (12). It is this variation in dose within the target volume which can be efficiency, but also which can induce the toxicity of interstitial brachytherapy. The linear quadratic model to calculate the biological equivalence of 2 Gy irradiation scheme most often hypofractionned, is theoretically applicable for doses per fraction less than 8 Gy. Nevertheless, the authors using the IPAS intra-operative (electrons, photons) apply this method of calculation for doses of 21 Gy in one fraction.

In our study, we propose to treat these patients with a total dose of 16 Gy in one fraction. This dose is calculated taking into account a report alpha/beta for the breast, on the order of 3.4 Gy for late toxicity and 4.6 Gy for local control (13). Applying the linear-quadratic model with alpha/beta for the breast of 4, 16 Gy in one fraction is calculated as radio-biologically equivalent to 53 Gy in conventional fractionation (14,15). Biological Equivalence of this dose is between the dose in the protocols IPAS intraoperative electron or X-ray photons of 50 kV (21 Gy in one fraction, 87 Gy EQD2 alpha/beta 4.6) (5.8) and the post-operative irradiation of 34-38 Gy in 10 fractions, 5 days (42 Gy EQD2 alpha/beta 4.6.

ELIGIBILITY:
Inclusion Criteria:

* Patient WITHinvasive breast cancer histologically proved: ductal, lobular, medullary, papillary, tubular or colloid:

  * All grades histo-prognostic
  * pT1 tumor size (<20 mm),
  * healthy Margins surgical
  * unifocal lesion
  * Any hormone receptor,
  * Any Her2 status,
  * No lymph node (sentinel lymphadenectomy or) or micrometastases (pN0, pN1mic)
* Age greater than or equal to 70 years
* Score Balducci I or II,
* Karnofsky index greater than or equal to 70%
* Time between lumpectomy and radiation less than 2 weeks
* Implementation of clips in the tumor bed intraoperatively,
* Patient having taken note of the information note and who signed the informed consent
* Patient receiving social security coverage.

Exclusion Criteria:

* Lobular carcinoma in situ or pure ductal carcinoma in situ or non-epithelial tumor type sarcoma or lymphoma,
* Component extensive ductal in situ associated
* Peritumoral lymphatic emboli,
* Distance Metastasis
* Inflammatory Breast Cancer,
* Multifocal tumor (covering a total distance inter-end of 40 mm or more)
* Previous treatment for this tumor including breast radiotherapy and / or chemotherapy neoadjuvant or adjuvant
* History of plastic surgery breast
* Unknown or safety margins positive for invasive carcinoma
* Absence of clips in the tumor bed,
* Time between lumpectomy and radiation greater than or equal to 2 weeks
* Active infection or other serious comorbidity that could prevent the patient receiving the treatment,
* History of cancer other than a basal cell skin or carcinoma in situ of the cervix or other cancer in complete remission for more than 5 years
* Psychiatric illness

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HANNOUN LEVI, Phd, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- [Derived] Hannoun-Levi JM, Cham Kee DL, Gal J, Schiappa R, Hannoun A, Gautier M, Boulahssass R, Peyrottes I, Barranger E, Ferrero JM, Chand ME, Doyen J. Accelerated partial breast irradiation for suitable elderly women using a single fraction of multicatheter interstitial high-dose-rate brachytherapy: Early results of the Single-Fraction Elderly Breast Irradiation (SiFEBI) Phase I/II trial. Brachytherapy. 2018 Mar-Apr;17(2):407-414. doi: 10.1016/j.brachy.2017.11.008. Epub 2017 Dec 15. PMID 29254856
- See also: Related Info — http://www.centreantoinelacassagne.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Irradiation and Accelerated Partial Breast (IPAS): Once the patient recorded in the trial, and after completion of a post-implant dosimetry scanner to analyze the dose distribution within the target volume and organs at risk, the patient is treated by irradiation and partial accelerated breast brachytherapy using high dose rate, delivering a total dose of 16 Gy in one fraction
  IPAS
Period: Overall Study
Arm/Group | Irradiation and Accelerated Partial Breast (IPAS)
Started | 31
Completed | 26
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- IPAS: Once the patient recorded in the trial, and after completion of a post-implant dosimetry scanner to analyze the dose distribution within the target volume and organs at risk, the patient is treated by irradiation and partial accelerated breast brachytherapy using high dose rate, delivering a total dose of 16 Gy in one fraction
  IPAS
Arm/Group | IPAS
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Region of Enrollment [Number; unit: participants]
  France | 37

OUTCOME MEASURES:

1. Primary Outcome: Rate of Acute Toxicity Within 180 Days of IPAS Mono Split Postoperatively in Patients Aged at Least of 70 Years With Breast Cancer at Low Risk of Local Recurrence (Low Risk Group of ESTRO IPAS Classification ESTRO)
Description: Rate of acute toxicity evaluated by a clinical examination, in consultation with the radiotherapist to 30, 90 days and 180 days.
  Common Toxicity Criteria classification for Adverse Events (CTCAE) in its fourth version is used.
Time Frame: 180 days
Measure: Number; unit: percentage of participants
Arm/Group | IPAS
Number analyzed (Participants) | 26
percentage of participants | 70

2. Secondary Outcome: Evaluation of the Quality of Life
Description: Analysis of the impact on self assessment by onco-geriatric aesthetic result evaluation Dosimetric data analysis in order to propose dose constraints for future inverse planning
Time Frame: 180 days
Reporting Status: Not Posted, anticipated posting 2021-11

ADVERSE EVENTS:
Arm/Group | IPAS
Serious Adverse Events (participants affected / at risk) | 3/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPAS (N=26)
left breast painful inflammatory syndroma (Reproductive system and breast disorders) | 1 (1)
tacchycardia (Cardiac disorders) | 1 (1)
right breast haematoma (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPAS (N=26)
BREAST FIBROSIS (Reproductive system and breast disorders) | 14 (14)
INJECTION SITE INFLAMMATION (Skin and subcutaneous tissue disorders) | 2 (2)
BREAST HAEMATOMA (Reproductive system and breast disorders) | 4 (4)
BREAST PAIN (Reproductive system and breast disorders) | 2 (2)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 5 (5)
RADIATION SKIN INJURY (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes